CLINICAL TRIAL: NCT05902611
Title: The Relationship Between Body Mass Index, Dental Eruption and Dental Caries Prevalence in School Children: A Cross-sectional, Observational Study
Brief Title: The Relationship Between Body Mass Index, Dental Eruption and Dental Caries Prevalence in School Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ibrahim Ahmed Hammad, Dentist, Al-Azhar University
Other Study IDs: 635/3505
Record Dates: First submitted 2023-06-03; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Body Mass Index; Dental Caries; Eruption
MeSH Terms: conditions — Dental Caries; Exanthema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: BMI determination, Eruption Time Assessment, Caries Assessment — BMI determination, Eruption Time Assessment, Caries Assessment

SUMMARY:
The aim of the current study will be to explore the relationship between body mass index, dental eruption and dental caries prevalence in school Children.

DETAILED DESCRIPTION:
Obesity is an abnormal accumulation of body fat. This accumulation of extra fat within the body may have either environmental or genetic causes . Obese children and adolescents are at increased risk for developing diabetes, metabolic problems, high blood pressure hypertension, coronary artery disease, sleep apnea, orthopedic problems, and psychosocial disorders.

Body mass index is the definition of obesity for children and adolescents. It is a formula that considers an individual's height and weight to determine body fat and health risk. For children it is calculated by this formula: weight ÷ (height x height).

For children and teens, BMI is age- and sex-specific and is often referred to as BMI-for-age. A child's weight status is determined using an age- and sex-specific percentile for BMI rather than the BMI categories used for adults. This is because children's body composition varies as they age and varies between boys and girls. Therefore, BMI levels among children and teens need to be expressed relative to other children of the same age and sex.

Obesity and dental caries are multifactorial conditions, both having comprehensive etiology and factors such as dietary habits and available nutrients, oral hygiene, or saliva . Changes in diet and lifestyle, such as an increase in wealth and access to carbohydrate-rich, high-calorie food and drinks could be attributed to the increase in the prevalence of both dental caries and obesity.

Several studies have evaluated the relationship between tooth decay and obesity; however, results are sometimes contradictory but recent studies showed that underweight children may experience higher dental caries than normal weight and overweight children.

Dental eruption is the emergence of the tooth into the oral cavity from its position in the alveolar crypt, and this process is influenced by genetic, systemic, general and local factors. It is positively related to the somatic growth (height and weight) of an individual.

Many studies worldwide describe how poor nutrition during the growth period adversely influences aspects of dental development, including delaying the eruption of deciduous and permanent teeth in underweight children than normal and overweight children. Postnatal growth and nutritional status have been linked to the eruption of primary teeth however; the studies assessing the association of obesity and permanent tooth development are few.

This complicated relation between oral health and body composition must be taken into consideration when treating children, hence the aim of this study is to identify if there is any relationship between dental caries and dental eruption with body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Parents and patients, acceptance and cooperation.
* children between 6 and 9 years of age.

Exclusion Criteria:

* Uncooperative child.
* Children with systemic disease that can affect their cooperation.

Ages: 6 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: The aim of this study is to find out the relationship between body mass index, dental eruption and dental caries in children aged 6 to 9 years, based on the previous study by Anu 2020 (15) who reported a correlation of -0.08 between body mass index and eruption status of permanent mandibular molar; a total sample size of 1224 will be sufficient with power 80 % and 5% significant level. The sample size was calculated by PASS 2008.
Sampling Method: Non-Probability Sample
Enrollment: 1224 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index using this equation: weight in kilograms divided by the square of height in meters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Nabil Abbas, PHD, Study Chair — Al-Azhar University
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Perez L, Irigoyen ME, Zepeda M. Dental caries, tooth eruption timing and obesity: a longitudinal study in a group of Mexican schoolchildren. Acta Odontol Scand. 2010 Jan;68(1):57-64. doi: 10.3109/00016350903449367. PMID 19958253
- See also: Related Info — https://systematicreviewsjournal.biomedcentral.com/articles/10.1186/2046-4053-1-57
- See also: Related Info — https://link.springer.com/article/10.1186/s12903-019-0950-y